CLINICAL TRIAL: NCT02912546
Title: Évaluation en IRM (séquence ASL) de la Variation de Perfusion cérébrale liée à la Position Corporelle.
Brief Title: Cerebral Perfusion Associated With Postural Changes: an ASL MR Perfusion Study
Acronym: PerfIRMAVC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Center of Martinique (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: 16/B/03
Record Dates: First submitted 2016-09-19; First posted 2016-09-23 (Estimated); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Brain Ischemia
Keywords: Stroke, Acute
MeSH Terms: conditions — Brain Ischemia; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Eighteen healthy subjects and eighteen hypertensive patients (men and women) will be enrolled. A 1.5 Tesla MRI device with a large magnet bore (70 cm) will be used, allowing positions change. Two measures will be performed, one in supine position and the other in head down position (-20°). A 3D FSE ASL sequence will be acquired and Cerebral Blood Flow (CBF) maps will be reconstructed. Volume of interest (VOI) will be placed on cortical grey matter (frontal and posterior gyrus), on subcortical deep grey matter (caudate nuclei, thalami) and subcortical white matter (semi oval centers). Differences in CBF values (in mL/100g/min) will be analyzed using SAS 9.3 software for Windows (SAS Institute, Cary North Carolina, USA).
  Interventions: Procedure: MRI
- Stroke patients (Active Comparator): Eighteen stroke patients (men and women) will be enrolled. A 1.5 Tesla MRI device with a large magnet bore (70 cm) will be used, allowing positions change. Two measures will be performed, one in supine position and the other in head down position (-20°). A 3D FSE ASL sequence will be acquired and Cerebral Blood Flow (CBF) maps will be reconstructed. Volume of interest (VOI) will be placed on cortical grey matter (frontal and posterior gyrus), on subcortical deep grey matter (caudate nuclei, thalami) and subcortical white matter (semi oval centers). Differences in CBF values (in mL/100g/min) will be analyzed using SAS 9.3 software for Windows (SAS Institute, Cary North Carolina, USA).
  Interventions: Procedure: MRI

INTERVENTIONS:
Procedure: MRI — A 1.5 Tesla MRI device with a large magnet bore (70 cm) allowing positions change will be used. Two measures will be performed, one in supine position and the other in head down position (-20°). A 3D FSE ASL sequence will be acquired and CBF maps reconstructed. Volume of interest (VOI) will be placed on cortical grey matter (frontal and posterior gyrus), on subcortical deep grey matter (caudate nuclei, thalami) and subcortical white matter (semi oval centers

SUMMARY:
Postural changes are commonly used as therapeutic maneuver to enhance or reduce cerebral perfusion. For instance, in acute stroke, the patient can be positioned in head down tilt position so as to increase perfusion of cerebral tissues perfusion. In During stroke and in hypertensive patients and during stroke, varying degrees a various loss of cerebral autoregulation is loss are usually observed. The aim of this study is to assess cerebral perfusion with ASL perfusion in human subjects in different conditions: healthy, hypertensive and stroke.

DETAILED DESCRIPTION:
Material and methods:

Eighteen stroke patients, eighteen hypertensive patients and eighteen healthy subjects (men and women) will be enrolled. The investigator will use a 1.5 Tesla MRI device with a large magnet bore (70 cm) allowing positions change. Two measures will be performed, one in supine position and the other in head down position (-20°). A 3D FSE ASL sequence will be acquired and Cerebral Blood Flow (CBF) maps will be reconstructed. Volume of interest (VOI) will be placed on cortical grey matter (frontal and posterior gyrus), on subcortical deep grey matter (caudate nuclei, thalami) and subcortical white matter (semi oval centers). Differences in CBF values (in mL/100g/min) will be analyzed using SAS 9.3 software for Windows (SAS Institute, Cary North Carolina, USA).

Expected results and hypothesis:

CBF is expected to significantly vary between the supine and head down positions. It is expected to at least increase in the head down position, for stroke patients. For healthy subjects and hypertensive patients, cerebral autoregulation may limit CBF increase although an increasing trend for CBF is expected.

ELIGIBILITY:
Inclusion Criteria:

1. Group of stroke patients:

   * Patients between 40 and 70 years old, male or female
   * With supratentorial ischemia in subacute phase (> H24)
   * Patients with a recent ischemic stroke with an intracranial hemodynamic unstable and kept lying with head down of about 30
   * Patient given free and informed consent to participate in research or a family representative
   * Patient insured under the French social security system
2. Control Group:

1- Group of patients with Hypertension.

* Patients between 40 and 70 years old, matched for age and sex to stroke patients.
* With a hypertension diagnosed since 10 years old.
* Hypertension defined as three recommendations (OMS 1999, ANAES 1997 JNC VI): blood pressure 140 and / or 90 mmHg found at several consultations.

  2- Group with healthy people.
* Healthy person between 30 and 70 years old, women and men. Healthy character will be defined on the basis of a physical examination (measurement of heart rate and blood pressure ) and an examination to determine the absence of endocrine pathology ... ) and the absence of drug outlet continuous.
* Person insured under the French social security system.
* Person who given free and informed his consent to participate in research or a family representative.
* Person who are not participating in another clinical study.

Exclusion Criteria:

* Patients aged under 40 years and 71 years and older for patients in groups of stroke patients and patients with hypertension
* Person under 30 years and 71 years and older for healthy people
* Person who refuses or family the participation in the study
* Person with heart antecedent or spinal disease
* Contraindications to the realization of a MRI (pacemaker, claustrophobia, metallic body may be mobilized).
* Person not insured under the French social security system,
* Pregnant women
* Persons under guardianship or curatorship
* Persons deprived of liberty by a judicial or administrative decision
* Persons who are participating in another clinical study

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2019-09-05 (Actual)

PRIMARY OUTCOMES:
The change in the value of the cerebral blood flow | up to 1 year
  The endpoint is the change in the value of the cerebral blood flow ( ml / 100g / min) depending on the switching position ( 0 ° and -20 °). This development will be assessed in different brain regions . In particular, it will be searched in excess of a threshold of significance .
  This will be accomplished independently by two experienced readers (knowing that the variation between and within road has been assessed) . If a significant difference between the two players, it will be made a consensual common measure.

CONTACTS AND LOCATIONS:
Overall Officials: Mehdi MM MEJDOUBI, PhD, Principal Investigator — CHU de Fort de France
Locations (1):
- Centre Hospitalier Universitaire de Martinique, Fort-de-France, Martinique

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chalela JA, Alsop DC, Gonzalez-Atavales JB, Maldjian JA, Kasner SE, Detre JA. Magnetic resonance perfusion imaging in acute ischemic stroke using continuous arterial spin labeling. Stroke. 2000 Mar;31(3):680-7. doi: 10.1161/01.str.31.3.680. PMID 10700504
- [Result] Lovell AT, Marshall AC, Elwell CE, Smith M, Goldstone JC. Changes in cerebral blood volume with changes in position in awake and anesthetized subjects. Anesth Analg. 2000 Feb;90(2):372-6. doi: 10.1097/00000539-200002000-00025. PMID 10648324